CLINICAL TRIAL: NCT04314323
Title: National Registry of Idiopathic Retroperitoneal Fibrosis in China
Brief Title: National Registry of IRPF in China
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Wen Zhang, Professor, Peking Union Medical College Hospital
Other Study IDs: IRPF group in China
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Idiopathic Retroperitoneal Fibrosis
Keywords: Registry; Cohort-study; Idiopathic retroperitoneal fibrosis；
MeSH Terms: conditions — Retroperitoneal Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples from IRPF patients will be saved for DNA extration and study.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to establish a nation-wide cohort study of idiopathic retroperitoneal fibrosis (IRPF) in China.

Methods: All the patients fulfilling diagnostic criteria of IRPF would be enrolled from multi-centers around China. A online database system has been established.

Endpoints: The primary endpoint is to investigate the clinical manifestations of Chinese IRPF patients; the secondary endpoints including the demographic features,laboratory characteristics, immunological tests, imaging and pathological features, in addition, the treatment and prognosis of the disease.

DETAILED DESCRIPTION:
This is a multicenter registry study of IRPF patients. Newly diagnosed IRPF patients will be recruited from all over the China. Inclusion criteria: patients with newly diagnosed IRPF will be recruited. Exclusion criteria: patients with secondary forms of retroperitoneal fibrosis or malignancy are excluded.

The data will be uploaded through the platform of Chinese Rheumatology Information Platform. Demographic data, initial symptoms, disease duration, history of allergy, and physical examination, organ involvements, laboratory findings, radiological and pathological results, as well as treatment, side effects will be recorded.

This study was approved by the Medical Ethics Committee of PUMCH (Beijing, China). All patients will sign informed consent.

Statistical Analysis: All parameters are described in the standard summary statistics, including mean, standard deviation, minimum, and maximum. All statistical analyses will be performed by SPSS.

Endpoints: The primary endpoint is to investigate the organ involvements of Chinese IRPF patients. The secondary endpoints include the demographic features,laboratory characteristics, immunological tests, imaging and pathological features, in addition, the treatment and prognosis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Conforming to the diagnostic criteria of IRPF;Definite IRPF must have the following characteristics: (1) The typical finding of Imaging shows retroperitoneal mass, surrounding the abdominal aorta and iliac arteries, with encasement of ureters and/or organ dysfunction; (2) Exclusion of disease progression after standard glucocorticoid treatment; and (3) histopathological findings shows a ﬁbrous tissue with signs of chronic inﬂammation. The inﬂammatory component is comprised of lymphocytes, plasma cells and macrophages. Neutrophils and granulomas are rare ﬁndings. Possible IRPF required (1) and (2), but without histopathological examination.

Exclusion Criteria:

* None of them met the criteria for other autoimmune diseases. None had malignant disease. Secondary forms of RPF related to drugs, infections, malignancies, Erdheim-Chester disease and IgG4-RD, need to be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: IRPF patients around China.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-03-17 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Organ involvements of Chinese IRPF patients | 5 years
  To calculate the percentage of organ involvements in at least 500 patients.

SECONDARY OUTCOMES:
Response rate of treatment with glucocorticoids and immunosuppressants on IRPF in China | 5 years
Relapse rate of IRPF patients in China | 5 years
The correlation between baseline disease activities and relapse rate. | 5 years
Ten year survival rate of patients with IRPF in China. | 10 years
The imaging features of involved organs. | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes